CLINICAL TRIAL: NCT01896713
Title: To Determine if MultiSpectral 3 Tesla MRI Can Provide Added Value in the Detection of Significant Cancers in Patients o n Active Surveillance for Prostate Cancer
Brief Title: The Value of MultiSpectral 3 Tesla MRI in Active Surveillance of Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Principal Investigator, Masoom Haider, Chief, Department of Medical Imaging, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 154-2009
Record Dates: First submitted 2013-01-07; First posted 2013-07-11 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; MRI; TRUSBx
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diagnostic: Single Arm (Other): Imaging (MS3TMRI)
  Interventions: Other: MS3TMRI

INTERVENTIONS:
Other: MS3TMRI — Multispectral 3 Tesla MRI imaging with contrast followed by biopsy
  Other Names: Multispectral 3 Tesla MRI imaging

SUMMARY:
MultiSpectral 3 Tesla MRI (MS3TMRI) can increase the yield of Trans Rectal Ultrasound Biopsy (TRUSBx) to improve identification of patients on active surveillance requiring treatment.

DETAILED DESCRIPTION:
This is a prospective single arm study. 120 patients at risk for significant occult prostate cancer on an active surveillance program will undergo MS3TMRI followed by a standard TRUSBx and additional biopsies guided by the MS3TMRI results. The positive predictive value (PPV) of MS3TMRI-TRUSBx for cancer requiring consideration of therapy will be compared to the PPV of TRUSBx alone. MS3TMRI consists of T2, diffusion-weighted imaging (DWI), dynamic contrast enhanced MRI (DCEMRI), proton MR spectroscopy (MRS) interpreted by a radiologist and by CAD methods validated on whole mount prostate specimens.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in active surveillance at Sunnybrook Health Sciences Centre, requiring biopsy as part of surveillance protocol.
* Clinically eligible for radical prostatectomy and willing to undergo surgery
* Clinically eligible for and willing to undergo ultrasound biopsy within 8 weeks of MRI

Exclusion Criteria:

* Claustrophobia
* Contraindication to MRI
* Contraindication to receiving low molecular weight MRI contrast agent
* Prior hormone therapy except 5-alpha reductase inhibitors such as Avodart. FloMax etc
* Clinically suspected or known compromised renal function or calculated estimated Glomerular Filtration Rate (eGFR) <30ml/min

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2010-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The Positive Predictive Value (PPV) of MS3TMRI-TRUSBx for detection of a patient with a cancer burden requiring consideration of immediate therapy. | The outcome measure will be evaluated at the time of the results of the TRUSbx which will be approximately 2 weeks after the biopsy
  Compare the targeted biopsy to the random biopsies

SECONDARY OUTCOMES:
The number of cores required for diagnosis of prostate cancer for MS3TMRI-TRUSBx versus TRUSBx alone | The outcome measure will be evaluated at the time of the results of the TRUSbx which will be approximately 2 weeks after the biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Masoom Haider, MD, Principal Investigator — Sunnybrook Health Sciences Centre, University of Toronto
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada